CLINICAL TRIAL: NCT04901715
Title: Functional Studies of Novel Genes Mutated in Primary Ciliary Dyskinesia II: Genotype to Phenotype
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20-3465; R01HL117836 (NIH)
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: Mucociliary clearance; Radial Spoke Head Component 1 (RSPH1); Dynein Axonemal Heavy Chain 5 (DNAH5); albuterol; short acting beta-adrenergic (SABA); SABA
MeSH Terms: conditions — Ciliary Motility Disorders | interventions — Albuterol; Nebulizers and Vaporizers; apaflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Genotypes associated mild phenotype (Active Comparator): Subjects with 2 confirmed mutations in RSPH1, Radial Spoke Head Component 9 (RSPH9), Radial Spoke Head Component 4A (RSPH4a), or Dynein Axonemal Heavy Chain 11 (DNAH11). This group may also include subjects with mutations in newly identified genes that are associated with a milder clinical phenotype.
  Interventions: Drug: Albuterol; Diagnostic Test: Technetium99m - Sulfur Colloid (Tc99m-SC)
- Genotypes associated with severe phenotype (Active Comparator): Subjects with 2 confirmed mutations in DNAH5, Dynein Axonemal Intermediate Chain 1 (DNAI1), Coiled-Coil Domain Containing 39 (CCDC39), or Coiled-Coil Domain Containing 40 (CCDC40). This group may also include subjects with mutations in newly identified genes that are associated with a more severe clinical phenotype.
  Interventions: Drug: Albuterol; Diagnostic Test: Technetium99m - Sulfur Colloid (Tc99m-SC)
- Healthy Control (Active Comparator): Healthy subjects with no pre-existing lung disease.
  Interventions: Drug: Albuterol; Diagnostic Test: Technetium99m - Sulfur Colloid (Tc99m-SC)

INTERVENTIONS:
Drug: Albuterol — Albuterol HFA Metered Dose Inhaler (90mcg/puff). Subjects to use 4 puffs one time.
  Other Names: ProAir HFA hydrofluoroalkane (HFA) Inhaler; Ventolin HFA (hydrofluoroalkane) Inhaler
Diagnostic Test: Technetium99m - Sulfur Colloid (Tc99m-SC) — Aerosolized radiolabeled Tc99m-sulfur colloid will be delivered using a modified Pari-LC Star nebulizer. The activity of Tc99m-SC loaded in the nebulizer will be adjusted to provide an estimated 40 microcurie (µCi) deposited in the lung for the MCC/CC scan. Patients between the age 12-18 years old will receive three quarters of the adult dose to account for the smaller lung volume.

SUMMARY:
The purpose of this study is to measure mucociliary clearance (MCC) in groups of subjects with the disease Primary Ciliary Dyskinesia (PCD) caused by mutations in different genes, and compare to healthy subjects. Some of these genes are associated with a milder clinical phenotype. This study seeks to determine if the milder phenotype is a result of mutations in a set of specific genes. The hypothesis is that subjects with PCD caused by mutations in the milder group will maintain a low, but significant rate of mucociliary clearance, while patients with mutations in genes in the more severe group will have a complete absence of mucociliary clearance. These studies will help inform future treatment strategies.

DETAILED DESCRIPTION:
Participants will undergo screening with basic physical exam and lung function testing at the start of the study. Participants will then inhale a radiolabeled substance and undergo medical imaging to measure the clearance of mucus in the airways. Albuterol will be administered after the first imaging is completed. Lung function testing will be repeated. Finally, medical imaging will be repeated two more times to further look at clearance of mucus in the lungs. The study will be completed in one day and will last about 6 hours.

ELIGIBILITY:
Inclusion Criteria for PCD Patients

* Confirmed PCD diagnosis with identified genetic mutations
* Negative pregnancy test for females who are not s/p hysterectomy with oophorectomy
* Forced Expiratory Volume (FEV1) of at least 30 percent of predicted

Inclusion Criteria for Healthy Controls:

* Age ≥ 18 years old
* Subjects must have an Forced vital capacity (FVC), Forced Expiratory Volume in one second (FEV1) and FVC/FEV1 of at least 80% of predicted.

Subjects who fall out of the normal range will be offered a copy of the test to share with their personal physician.

* No pre-existing lung disease (asthma, cystic fibrosis, etc.).
* Negative pregnancy test for females who are not s/p hysterectomy with oophorectomy.

Exclusion Criteria:

* Any chronic medical condition considered by the PI as a contraindication to the exposure study including significant cardiovascular disease, diabetes, chronic renal disease, chronic thyroid disease, immunodeficiency, history of tuberculosis
* Any acute infection requiring antibiotics within 4 weeks of study.
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
* Medications which may impact the results of the study treatment, or may interfere with any other medications potentially used in the study (to include steroids, beta antagonists, non-steroidal anti-inflammatory agents)
* Active smoking to include e-cigarettes within 1 year of the study, or lifetime of > 10 pack years of smoking
* History of vaping or current vaping.
* Viral upper respiratory tract infection within 4 weeks of challenge.
* Radiation exposure history in the past year which would be outside the safe levels
* Pregnant or lactating women will also be excluded since the risks associated with radiation are unknown and cannot be justified
* Use of the following medications:

  1. Use of beta blocking medications
  2. Receipt of Live Attenuated Influenza Vaccine (LAIV), also known as FluMist , within the prior 30 days, or any vaccine within the prior 5 days
  3. Multivitamins, Vitamin C or E or herbal medications in the 4 days prior to the treatment visit
  4. Non-steroidal anti-inflammatory drugs in the 4 days prior to the treatment visit.
* Allergy/sensitivity to study drugs or their formulations:
* Known Immunoglobulin E (IgE) mediated hypersensitivity to albuterol
* Physical/laboratory indications:

  1. Temperature > 37.8 degrees Celsius (C)
  2. Subjects >15 years- Systolic BP >150 mm hg or < 90 mm Hg or diastolic BP> 90 mm Hg or < 50 and Subjects 12-15 years - Systolic BP > 130 mmHg or < 80 mmHg or diastolic BP > 80 or <40
  3. Oxygen saturation of < 93 percent
* Inability or unwillingness of a participant to give written informed consent.

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Ostrowski, PhD, Principal Investigator — University of North Carolina at Chapel Hil
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: 12-36 months following publication
Access Criteria: Investigators with IRB, IEC, or REB approval and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 27 participants who signed informed consent, three participants failed screening and were ineligible to continue participation and did not receive the study intervention.
Groups:
- Genotypes Associated With Mild Phenotype: Subjects with 2 confirmed mutations in Radial Spoke Head Component 1 (RSPH1), Radial Spoke Head Component 9 (RSPH9), Radial Spoke Head Component 4A (RSPH4a), or Dynein Axonemal Heavy Chain 11 (DNAH11). This group may also include subjects with mutations in newly identified genes that are associated with a milder clinical phenotype.
  Albuterol: Albuterol HFA hydrofluoroalkane (HFA) Metered Dose Inhaler (90mcg/puff). Subjects to use 4 puffs one time.
  Technetium99m - Sulfur Colloid (Tc99m-SC): Aerosolized radiolabeled Tc99m-sulfur colloid will be delivered using a modified Pari-LC Star nebulizer. The activity of Tc99m-SC loaded in the nebulizer will be adjusted to provide an estimated 40 microcurie (µCi) deposited in the lung for the mucociliary clearance cough clearance (MCC/CC) scan. Patients between the age 12-18 years old will receive three quarters of the adult dose to account for the smaller lung volume.
- Healthy Control: Healthy subjects with no pre-existing lung disease.
  Albuterol: Albuterol HFA Metered Dose Inhaler (90mcg/puff). Subjects to use 4 puffs one time.
  Technetium99m - Sulfur Colloid (Tc99m-SC): Aerosolized radiolabeled Tc99m-sulfur colloid will be delivered using a modified Pari-LC Star nebulizer. The activity of Tc99m-SC loaded in the nebulizer will be adjusted to provide an estimated 40 microcurie (µCi) deposited in the lung for the MCC/CC scan. Patients between the age 12-18 years old will receive ¾ of the adult dose to account for the smaller lung volume.
Period: Overall Study
Arm/Group | Genotypes Associated With Mild Phenotype | Genotypes Associated With Severe Phenotype | Healthy Control
Started | 10 | 8 | 9
Completed | 8 | 8 | 8
Not Completed | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Genotypes Associated With Mild Phenotype: Subjects with 2 confirmed mutations in RSPH1, Radial Spoke Head Component 9 (RSPH9), Radial Spoke Head Component 4A (RSPH4a), or Dynein Axonemal Heavy Chain 11 (DNAH11). This group may also include subjects with mutations in newly identified genes that are associated with a milder clinical phenotype.
  Albuterol: Albuterol HFA Metered Dose Inhaler (90mcg/puff). Subjects to use 4 puffs one time.
  Technetium99m - Sulfur Colloid (Tc99m-SC): Aerosolized radiolabeled Tc99m-sulfur colloid will be delivered using a modified Pari-LC Star nebulizer. The activity of Tc99m-SC loaded in the nebulizer will be adjusted to provide an estimated 40 microcurie (µCi) deposited in the lung for the MCC/CC scan. Patients between the age 12-18 years old will receive ¾ of the adult dose to account for the smaller lung volume.
- Genotypes Associated With Severe Phenotype: Subjects with 2 confirmed mutations in DNAH5, Dynein Axonemal Intermediate Chain 1 (DNAI1), Coiled-Coil Domain Containing 39 (CCDC39), or Coiled-Coil Domain Containing 40 (CCDC40). This group may also include subjects with mutations in newly identified genes that are associated with a more severe clinical phenotype.
  Albuterol: Albuterol HFA Metered Dose Inhaler (90mcg/puff). Subjects to use 4 puffs one time.
  Technetium99m - Sulfur Colloid (Tc99m-SC): Aerosolized radiolabeled Tc99m-sulfur colloid will be delivered using a modified Pari-LC Star nebulizer. The activity of Tc99m-SC loaded in the nebulizer will be adjusted to provide an estimated 40 microcurie (µCi) deposited in the lung for the MCC/CC scan. Patients between the age 12-18 years old will receive ¾ of the adult dose to account for the smaller lung volume.
- Total: Total of all reporting groups
Arm/Group | Genotypes Associated With Mild Phenotype | Genotypes Associated With Severe Phenotype | Healthy Control | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 0 | 6
  Between 18 and 65 years | 4 | 5 | 8 | 17
  >=65 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 3 | 9
  Male | 3 | 7 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 7 | 8 | 6 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 8 | 8 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Baseline MCC (Ave60Clr; Average Clearance Over 60 Minutes)
Description: The average percent clearance in subjects with Primary Ciliary Dyskinesia (PCD) caused by mutations associated with mild and severe clinical phenotypes. Prior to each MCC study, a transmission Co57 scan will be performed to define the lung boundaries, to assign regions of interest, and to normalize these regions for lung volume differences. Radiolabeled Tc99m-sulfur colloid will be delivered using a modified Pari-LC Star nebulizer. The subject will then (within a minute of final inhalation maneuver) be seated in front of a large-field-of-view gamma camera to begin acquiring consecutive 2 minute images. The first two-2-minute images will provide initial, time zero activity (i.e. 100% retention) followed by the same imaging at the start of every 10-minute period until 1 hour has passed to assess baseline MCC. Clearance will be determined by measuring the decrease in radiolabeled Tc99m-sulfur colloid in the lungs over time.
Time Frame: 60 minutes
Population: One participant was originally included in the Genotypes Associated with Mild Phenotype Arm based on available knowledge. Upon further study of the genotype, it was concluded that this participant did not meet the criteria for a mild phenotype and was therefore excluded from the analysis.
Measure: Median (Inter-Quartile Range); unit: percent clearance
Arm/Group | Genotypes Associated With Mild Phenotype | Genotypes Associated With Severe Phenotype | Healthy Control
Number analyzed (Participants) | 7 | 8 | 8
percent clearance | 1.4 [-0.42 to 2.60] | -1.1 [-1.30 to 2.70] | 7.3 [4.9 to 9.1]
Statistical Analysis 1: Comparison: Genotypes Associated With Severe Phenotype vs Healthy Control; Test type: Other; p = 0.002, ANOVA
Statistical Analysis 2: Comparison: Genotypes Associated With Mild Phenotype vs Healthy Control; Test type: Other; p = 0.054, ANOVA
Statistical Analysis 3: Comparison: Genotypes Associated With Mild Phenotype vs Genotypes Associated With Severe Phenotype; Test type: Other; p = 0.27, ANOVA

2. Secondary Outcome: Change in MCC (Ave120Clr-Ave60Clr;Average Clearance Between 60 and 120 Minutes)
Description: The change in average percent clearance after the administration of albuterol in subjects with PCD caused by mutations associated with mild and severe clinical phenotypes PCD patients with mild disease compared to PCD patients with more severe disease. A transmission Cobalt57 scan will be performed to define the lung boundaries. Radiolabeled Tc99m-sulfur colloid (Technetium99m) will be delivered using a modified nebulizer. The subject will be seated in front of a large-field-of-view gamma camera to begin consecutive 2 minute images. The first two-2-minute images will provide initial, time zero activity followed by the same imaging at every 10-minute period until 1 hour. Subjects will then inhale 4 puffs of albuterol from the Metered Dose Inhaler (MDI) and consecutive 2 minute imaging continues for the next hour to assess the effect of albuterol on MCC. Clearance will be determined by measuring the decrease in radiolabeled Tc99m-sulfur colloid in the lungs over time.
Time Frame: 120 minutes
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent clearance
Arm/Group | Genotypes Associated With Mild Phenotype | Genotypes Associated With Severe Phenotype | Healthy Control
Number analyzed (Participants) | 7 | 8 | 8
percent clearance | 0.82 [-0.53 to 1.90] | -0.42 [-1.40 to 2.50] | 9.7 [1.82 to 12.00]
Statistical Analysis 1: Comparison: Genotypes Associated With Severe Phenotype vs Healthy Control; Test type: Other; p = 0.014, ANOVA
Statistical Analysis 2: Comparison: Genotypes Associated With Mild Phenotype vs Healthy Control; Test type: Other; p = 0.066, ANOVA
Statistical Analysis 3: Comparison: Genotypes Associated With Mild Phenotype vs Genotypes Associated With Severe Phenotype; Test type: Other; p = 0.58, ANOVA

3. Other Pre Specified Outcome: Change in Cough Clearance (Ave150Clr-Ave120Clr; Average Clearance Between 120 and 150 Minutes)
Description: The change in average percent of cough clearance in subjects with PCD caused by mutations associated with mild and severe clinical phenotypes PCD patients with mild disease compared to PCD patients with more severe disease.
  After completion of baseline MCC measurement and post-Albuterol MCC measurement. Subjects will cough a total of 30 times over a 30-minute period to assess cough clearance by gamma imaging over that period. Clearance will be determined by measuring the decrease in radiolabeled Tc99m-sulfur colloid in the lungs over time.
Time Frame: 150 minutes
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through 96 hours after completion of the single 8-hour study visit.
Arm/Group | Genotypes Associated With Mild Phenotype | Genotypes Associated With Severe Phenotype | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT04901715/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT04901715/ICF_001.pdf